CLINICAL TRIAL: NCT00131846
Title: Effect of Low Dose Thiazide Diuretics on New Onset Type 2 Diabetes in Patients With Essential Hypertension
Brief Title: Diuretics In the Management of Essential Hypertension (DIME) Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kyoto University (Other)
Collaborators: University of the Ryukyus (Other)
Responsible Party: Principal Investigator, Takeshi Morimoto, Professor of Medicine, Kyoto University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H15-choju-003
Record Dates: First submitted 2005-08-17; First posted 2005-08-19 (Estimated); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Hypertension
Keywords: Thiazide diuretics; Essential hypertension; Type 2 diabetes; Randomized clinical trial; Cost-effectiveness
MeSH Terms: conditions — Hypertension; Essential Hypertension; Diabetes Mellitus, Type 2 | interventions — Sodium Chloride Symporter Inhibitors

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Diuretics use
  Interventions: Drug: Thiazide diuretics
- 2 (Active Comparator): No diuretics use
  Interventions: Drug: No diuretics

INTERVENTIONS:
Drug: Thiazide diuretics — Any dosage, frequency, and duration
  Arms: 1
Drug: No diuretics — Any antihypertensive regimen other than diuretics
  Arms: 2

SUMMARY:
The purpose of DIME is to evaluate the safety (i.e. new onset of diabetes and other metabolic adverse events), efficacy and cost-effectiveness of antihypertensive treatment with low dose diuretics. The researchers' hypothesis is that use of low dose thiazide diuretics is metabolically safe when used with other appropriate antihypertensives, effective in reduction of blood pressure and cheaper than treatment without diuretics. Therefore, this study is an equivalence trial.

DETAILED DESCRIPTION:
There has been substantial evidence from clinical trials to support the rationale of use of thiazide diuretics in patients with essential hypertension. Diuretics may be more effective in reduction of blood pressure in Japanese patients than Caucasian because of higher salt intake. Moreover, given a large number of hypertensive population here, diuretics may be the most cost-effective antihypertensive agent. Japanese physicians, however, tend to avoid diuretics even in elderly hypertensive patients because of much concern over metabolic adverse events including new onset diabetes, which is deemed to increase cardiovascular risk. Although it is unlikely that use of low dose (12.5 mg of HCTZ or less) diuretics is associated with metabolic adverse events when they are given with any other appropriate antihypertensive agents (e.g. Ca antagonist, ACE inhibitor, ARB, K sparing diuretics) other than β-blockers, the researchers have to confirm the safety of low dose diuretics in terms of new onset diabetes in Japanese, who are assumed to be "diabetes prone" based upon thrifty gene hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Aged 30 to 79 years
* With blood pressure being >150/>90 if they are not on any antihypertensive treatment
* With blood pressure being >140/>90 if they are already on antihypertensive drugs
* No history of type 2 diabetes
* No history of gout

Exclusion Criteria:

* With supine blood pressure being >200/>120
* Patients already on antihypertensive treatment if duration of treatment and drugs used are not identified
* Patients already on thiazide diuretics
* With type 2 diabetes
* With gout or hyperuricaemia (>8.0 mg/dl)
* With hypokalemia（<3.5mmol/L）
* With erectile dysfunction
* With renal dysfunction (s-creatinine > 2.0 mg/dL)
* With history of serious adverse reaction to thiazide diuretics
* With history of stroke or myocardial infarction within 6 months
* With history of percutaneous coronary intervention (PCI) or coronary artery bypass graft (CABG) within 6 months or in whom these interventions are planned
* With heart failure or left ventricular dysfunction (ejection fraction<40%)
* Patients who should be on thiazide diuretics
* With history of malignant tumor within 5 years
* Pregnant, possibility of pregnancy, or during breast feeding
* Patients who are deemed not eligible for this study for any reason

Ages: 30 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1130 (Actual)
Dates: Start 2004-04 (Actual); Primary Completion 2012-08 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
New onset type 2 diabetes (WHO criteria 1998) | five years

SECONDARY OUTCOMES:
Treatment resistant hypokalemia less than 3.5mEq/L | five years
Ischemic and hemorrhagic Strokes excluding transient ischemic attacks and secondary causes | five years
Myocardial infarction | five years
Hospitalization due to heart failure | five years
Arteriosclerosis obliterans (ASO) | five years
Total death | five years
Blood pressure | five years
Lipid profile | five years
HbA1c | five years
Fasting blood sugar | five years
Direct Cost | five years
Gout (American College of Rheumatology 1997 criteria C) | five years

CONTACTS AND LOCATIONS:
Overall Officials: Shinichiro Ueda, MB, ChB, PhD, Principal Investigator — Department of Clinical Pharmacology & Therapeutics, University of the Ryukyus
Locations (1):
- University of the Ryukyus, Nishihara, Okinawa, Japan

REFERENCES:
- [Derived] Ueda S, Morimoto T, Ando S, Takishita S, Kawano Y, Shimamoto K, Ogihara T, Saruta T; DIME Investigators. A randomised controlled trial for the evaluation of risk for type 2 diabetes in hypertensive patients receiving thiazide diuretics: Diuretics In the Management of Essential hypertension (DIME) study. BMJ Open. 2014 Jul 16;4(7):e004576. doi: 10.1136/bmjopen-2013-004576. PMID 25031188